CLINICAL TRIAL: NCT04906941
Title: Assessment of the Impact of Gadolinium Injection on the Measurement of the QSM Signal
Acronym: GADO-QSM
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JSY_2021_14
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: White Matter Disease
MeSH Terms: conditions — Leukoencephalopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — SWI QSM 1.0iso 8 echos sequence performed before and after the injected MRI prescribed as part of the treatment.
  * Sense 2 * 2: 9min33s

SUMMARY:
Patients meeting the inclusion and non-inclusion criteria will be offered to participate in the study. If they agree, they will perform an MRI without injection to obtain the QSM then perform the MRI with injection that was prescribed to them as part of the care, then they will perform a second time the MRI without injection to obtain the QSM. They will also answer a short questionnaire documenting their previous exposure to gadolinium.

DETAILED DESCRIPTION:
Patients meeting the inclusion and non-inclusion criteria will be offered to participate in the study. If they agree, they will perform an MRI without injection to obtain the QSM then perform the MRI with injection that was prescribed to them as part of the care, then they will perform a second time the MRI without injection to obtain the QSM. They will also answer a short questionnaire documenting their previous exposure to gadolinium.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* with an inflammatory CNS pathology
* to benefit as part of care from an MRI with injection of gadolinium
* consent to participate in the study
* beneficiary of a social protection scheme

Exclusion Criteria:

* pregnant or breastfeeding woman
* patient benefiting from a legal protection measure
* Patient having performed more than 3 MRI exams with gadolinium injection during his life

Secondary exclusion criteria :

* motion artifact not allowing image interpretation
* patient who has not completed one of the following sequences: T1 anatomical, FLAIR, or QSM pre-gadolinium injection.

Secondarily excluded patients will be replaced up to a maximum of 25 patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting the inclusion and non-inclusion criteria will be offered to participate in the study. If they agree, they will perform an MRI without injection to obtain the QSM then perform the MRI with injection that was prescribed to them as part of the care, then they will perform a second time the MRI without injection to obtain the QSM. They will also answer a short questionnaire documenting their previous exposure to gadolinium.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
mean of the delta observed between the QSM of the white matter before and after injection of gadolinium | 1 DAY
  mean of the delta observed between the QSM of the white matter before and after injection of gadolinium

CONTACTS AND LOCATIONS:
Locations (1):
- Hhopital fondation adolphe de rothschild, Paris, Paris, France